CLINICAL TRIAL: NCT05214820
Title: Clinical Assessment of the Therapeutic Potential of 177Lu-PSMA Endoradiotherapy for the Treatment of Upper Metastatic Gastric Cancers Using 68Ga-PSMA PET-based Dosimetry
Brief Title: 68Ga-PSMA PET Imaging of Upper Metastatic Gastric Cancers to Determine Eligibility to Endoradiotherapy
Acronym: ERD2021
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-4378
Record Dates: First submitted 2021-12-09; First posted 2022-01-31 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Upper Digestive Tract Cancer
Keywords: Imaging; 68Ga-PSMA; Dosimetry; Positron emission tomography (PET)

STUDY DESIGN:
Intervention Model Description: Prospective pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm with 68Ga-PSMA (Experimental): All participants will undergo a PET scan with 68Ga-PSMA
  Interventions: Biological: Radiopharmaceutical 68Ga-PSMA

INTERVENTIONS:
Biological: Radiopharmaceutical 68Ga-PSMA — Injection of 68Ga-PSMA followed by 3 PET/CT acquisitions

SUMMARY:
Upper gastrointestinal (GI) cancers are a major health problem in Canada. At the metastatic stage, options are limited (usually chemotherapy, immunotherapy, personalized therapies under research protocols). These options are not applicable to all patients and may have significant toxicities. Endoradiotherapy (ERT) using a radioisotope coupled with a localization vector specifically targeting tumor cells to deliver a localized dose of radiation therapy is a promising avenue as it can treat disseminated neoplastic disease in a specific manner sparing healthy tissue with minimal side effects. The main goal of this study is to confirm that patients with upper GI cancer would be eligible for ERT (177Lu-PSMA treatment by using 68Ga-PSMA PET/CT assessment).

DETAILED DESCRIPTION:
Background: Upper gastrointestinal (GI) cancers are a major health problem in Canada. At the metastatic stage, options are limited (usually chemotherapy, immunotherapy, personalized therapies under research protocols). These options are not applicable to all patients and may have significant toxicities. Endoradiotherapy (ERT) using a radioisotope coupled with a localization vector specifically targeting tumor cells to deliver a localized dose of radiation therapy is a promising avenue as it can treat disseminated neoplastic disease in a specific manner sparing healthy tissue with minimal side effects.

177Lu-PSMA would be a potentially usable ERT agent for upper GI cancers. Initially developed for prostate cancer, for which it has been successfully proven, it targets the PSMA protein found on tumor cells or their microenvironment. Its localization is usually confirmed by imaging with 68Ga-PSMA, which is the other component of its theranostic pair.

There are many case reports showing significant accumulation of 68Ga-PSMA in upper GI cancers, but there are no prospective studies to determine with certainty whether these are isolated cases or whether these tumors consistently uptake this agent; the same uptake that determines whether 177Lu-PSMA ERT has potential efficacy for these patients.

We believe that 177Lu-PSMA ERT could provide an effective radiation dose to treat metastatic high-grade GI cancers without exceeding acceptable dose limits to healthy tissue, providing a new therapeutic avenue for this patient group.

Objective:

1. To confirm that patients with upper gastric cancers would be eligible for 177Lu-PSMA treatment by using 68Ga-PSMA PET/CT assessment, according to the criteria suggested by the European Association of Nuclear Medicine (EANM) (tumor uptake 1.5 times higher than the liver)
2. Determine tumor heterogeneity (proportion of tumor lesions identified by computed tomography (CT) that capture 68Ga-PSMA) in each patient;
3. Determine the proportion of patients with lesions that do not accumulate 68Ga-PSMA;
4. Calculate the pharmacokinetics of 68Ga-PSMA by serial PET imaging;
5. Calculate dosimetry of healthy and tumor tissues;

Study population: Adults with upper metastatic gastric cancer (adenocarcinomas of the esophagus, stomach, bile ducts and pancreas)

Procedure and Follow-up: Patient will undergo 68Ga-PSMA PET imaging at different post-injection times (total visit duration of approximately half a day). Clinical data will be collected from this imaging and from the participant's medical record (demographic, treatment, medication, pathology, lab test results) for a 2-year follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Active cancer of the type adenocarcinoma (of the esophagus, of the stomach, of the bile ducts, or of the pancreas) documented by a CT scan performed within the last 8 weeks at the time of recruitment.

  * An active cancer is defined as at least one lesion identified as stable or progressive neoplastic on CT imaging.
  * A lesion treated with local therapy (e.g., external radiotherapy, cryoablation, radiofrequency ablation, resection) is not counted for inclusion criteria if this is done between the CT scan and the 68Ga-PSMA PET imaging. A lesion treated prior to the last CT scan may be considered eligible if progression is documented at the last CT scan.
* Able to provide free and informed consent.
* Feasibility to perform 68Ga-PSMA PET within 2 months of the CT scan that was used for inclusion.

Exclusion Criteria:

* Other active cancer (non-metastatic non-melanoma skin cancer excluded). Cancer in remission for at least 3 years will not be considered active.
* ECOG > 3.
* Pregnant woman.
* Unable to follow study rules.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-01-17 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Tumor uptake of 68Ga-PSMA | At 1 hour post-injection acquisition
  Proportion of participants with tumor uptake equal to or greater than 1.5 times the mean hepatic uptake (SUVmean) on 68Ga-PSMA PET according to the criteria suggested by the European Association of Nuclear Medicine (EANM)

SECONDARY OUTCOMES:
Tumor heterogeneity | At 1 hour post-injection acquisition
  Proportion of tumor lesions identified on CT that accumulate 68Ga-PSMA in each participant
Tumor lesions that do not accumulate 68Ga-PSMA | At 1 hour post-injection acquisition
  Proportion of patients with CT-identified tumor lesions that do not accumulate 68Ga-PSMA
Effective half-life of 68Ga-PSMA | At 30 minutes, 60 minutes and, 120 minutes post-injection
  Comparison of uptakes of 68Ga-PSMA in tumor lesions and healthy tissue at each time points
Radiation dose (mGy) | At 30 minutes, 60 minutes and120 minutes post-injection
  Estimated radiation dose (mGy) delivered to healthy and tumor tissues from 177Lu-PSMA extrapolated from 68Ga-PSMA results

CONTACTS AND LOCATIONS:
Locations (1):
- CIUSSS de l'Estrie- CHUS Hospital, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No